CLINICAL TRIAL: NCT05237882
Title: Internet-delivered CBT for Functional Gastrointestinal Disorders (FGID) in Youth - A Single Case Experimental Design Study Embedded in The Danish FGID Treatment Study
Brief Title: Internet-delivered CBT for Functional Gastrointestinal Disorders (FGID) in Youth: a Single Case Experimental Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Skovslund Nielsen, PhD-Student, Medical doctor, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGID Single case
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: A non-concurrent multi-variate baseline single-case experimental design (SCED) including 6 children and 6 adolescents with their parents. Baseline periods randomized between 5-15 days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children and Adolescents (Experimental): 6 children aged 8-12 years old, 6 adolescents aged 13-17 years old, fulfilling inclusion criteria will be included
  Interventions: Other: Internet delivered cognitive behavioural therapy for functional gastrointestinal disorders

INTERVENTIONS:
Other: Internet delivered cognitive behavioural therapy for functional gastrointestinal disorders — The offered treatment will be the Danish versions of the Swedish i-CBT programs for children. The child i-CBT program consists of 10 modules for the child and 10 for parents. The adolescent i-CBT program consists of 10 modules for the adolescent and 5 modules for the parents. Child and adolescents modules compose of exposure exercises for symptoms, behavioural analyses and affect labelling and are adjusted for the specific age group. Parent modules aim at supporting parents in helping their child to engage in the challenging exposure exercises. The family needs to select one parent to participate in the parent program. The participants will be expected to use approximately 4 hours per week. The programs will be delivered over ten weeks, and therapist support will be provided on a weekly basis.

SUMMARY:
Functional gastrointestinal disorders (FGID) are common among children and adolescents. They affect quality of life, cause functional disability, school absence and high health care use. Despite this there is a lack in treatment options.

The aim of the current study, embedded in The Danish FGID Treatment Study, is to investigate the detailed course of efficacy of Danish versions of Swedish Internet based cognitive behavioural therapy (i-CBT) programs for children and adolescents with FGID in a Danish clinical context. This will be done using a single case design study. Along with this, the impact of parental illness worries will be investigated.

DETAILED DESCRIPTION:
A non-concurrent multi-variate baseline single-case experimental design study (SCED) will be conducted. It will consist of a baseline phase, a treatment phase and a follow up phase, including 6 children and 6 adolescents with their parents.

Participants will be randomly assigned to a baseline length with a duration between 5-15 days.

The design, using a multi-variate baseline, enables each participant to form their own control as outcomes during the baseline are compared with outcomes during treatment. This means that if treatment is effectual a change in outcome measures will show during the treatment period no matter when the treatment period was started.

Outcome will be assessed daily from baseline to end of treatment using electronic self-report questionnaire, with a last, one week long, daily assessment at 3-month follow-up.

The questionnaire is designed for this specific study and consist of 8 items (modified to a daily question) from validated questionnaires, the scale is changed to an 11 point scale from 0(not at all) to 10(all the time) Outcome are: abdominal symptoms (2 items from PedsQL Gastro 9 items questionnaire), symptom catastrophizing (2 items from Visceral Short sensitivity Index questionnaire), avoidance and control behavior (2 items from IBS Behavioural Response Questionnaire), and symptom acceptance(2 items from Chronic Pain Acceptance Questionnaire for Adolescents 8-items)

In addition, a more comprehensive battery of questionnaires will be completed by the children and adolescents and the parent, respectively, at baseline, mid-treatment, end of treatment and at 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* child age: 8-12 years, adolescents: 13 - 17 years
* A primary diagnosis according to the ROME-IV criteria of one of the FGID sub-types: Irritable bowel syndrome (IBS) or functional abdominal pain not-otherwise-specified (FAP-NOS)
* The diagnosis should be documented by their regular physician in the somatic setting, and recommended routine medical investigations should be evaluated as normal or without clinical significance (include growth; blood samples including TSH, total IgA, IgA tissue transglutaminase, complete blood count, C-reactive protein analysis, liver enzymes; and fecal calprotectin)
* Stable dosage of FGID-related medication such as laxatives, anti-diarreal medication or pain-modulating psychopharmacological medication during the past month.

Exclusion Criteria:

* Another disease that explains the symptoms;
* Severe psychiatric or social problems (e.g., high level of suicidal ideation or ongoing abuse);
* Ongoing psychological treatment;
* Insufficient language or computer skills (patients and parents);
* Severe family problems (e.g. child abuse, parental substance abuse or severe psychiatric illness, ongoing custody fight)
* School absence of more than 40% over the past month.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Single Case Design Outcome: Change in gastrointestinal symptoms measured via Daily Items as part of self-report SCED-Questionnaire | Everyday during baseline (5-15 days before treatment start) and treatment (10 weeks) and during one week at 3 months follow-up
  The SCED-Questionnaire consists of 8 daily items about Gastrointestinal symptoms, catastrophizing, Avoidance and control, acceptance. Answered on a 11 point scale from 0 ("not at all") to 10 ("all the time")
Change in gastrointestinal symptoms assessed by PedsQL Gastro Symptom Scales | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The self-report questionnaire revised version of PedsQL Gastro Symptom Scales, with 9 items. Answered on a 5 point scale from 0 ("never") to 4 ("almost always)
Change in gastrointestinal symptoms rated by parents assessed by PedsQL Gastro Symptom Scales | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The parent-report questionnaire revised version of PedsQL Gastro Symptom Scales, with 9 items. Answered on a 5 point scale from 0 ("never") to 4 ("almost always)

SECONDARY OUTCOMES:
Single Case Design Outcome: Change in catastrophizing, avoidance and control and acceptance via Daily Items, measured as part of self-report SCED-Questionnaire | Everyday during baseline (5-15 days before treatment start) and treatment (10 weeks) and during one week at 3 months follow-up
  Measured as part of self-report SCED-Questionnaire of 8 daily items about Gastrointestinal symptoms, catastrophizing, Avoidance and control, acceptance. Answered on a 11 point scale from 0 ("not at all") to 10 ("all the time")
Changes in Quality of life assessed by the Pediatric Quality of Life Inventory | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The self-report questionnaire Pediatric Quality of Life Inventory 8-12-year version for children, 13-18-year version for adolescents. 23 items, Answered on a 5 point scale from 0 ("never") to 4 ("almost always)
Changes in Quality of life rated by parents assessed by Pediatric Quality of Life Inventory | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The parent-report questionnaire Pediatric Quality of Life Inventory for parents, (Parent report for children aged 8-12 years, and parent report for adolescents aged 13-17 years) . 23 items, Answered on a 5 point scale from 0 ("never") to 4 ("almost always)
Changes in Pain intensity measured by the self-report rating scale, Faces pain scale, revised | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The scale consists of 6 faces representing least to most pain, and each face is connected to a number from 0 (no pain) - 10 (most pain),
Changes in Pain intensity rated by parents Measured by the parent-report rating scale, Faces pain scale, revised. | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The scale consists of 6 faces representing least to most pain, and each face is connected to a number from 0 (no pain) - 10 (most pain),
Changes in Overall symptom load measured by the self-report questionnaire Children somatization inventory , short (CSI) | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The questionnaire consist of 24 items Answered on a 5 point scale from 0 ("not at all") to 4 ("a whole lot")
Changes in Overall symptom load rated by parents measured by the parent-report questionnaire Children somatization inventory (parent report), short | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The questionnaire consists of 24 items Answered on a 5 point scale from 0 ("not at all") to 4 ("a whole lot")
Changes in Depression symptoms measured by the self-report questionnaire Mood and Feelings Questionnaire short | At baseline, after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The questionnaire consists of 13 items, answered on a 3 point scale: not true / sometimes true / true
Changes in General Anxiety symptoms measured by the self- report questionnaire Spence Children Anxiety Scale short | At baseline, after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  A 19 item-questionnaire answered on a 4 point scale from 0(never) to 3 (always)
Changes in General Anxiety rated by parents, Measured by the parent- report questionnaire Spence Children Anxiety Scale short, parent report | At baseline, after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  a19 item-questionnaire answered on a 4 point scale from 0(never) to 3 (always)
Changes in Specific Gastrointestinal Anxiety, Measured by the self-report questionnaire Visceral Sensitivity Index - Short | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  A 7 item-questionnaire answered on a 5 point scale from 0 (don't agree at all) to 5 (totally agree)
Changes in Avoidance and control behaviour measured by the self-report questionnaire irritable bowel syndrome-behavioural response questionnaire | At baseline, mid-treatment, end-treatment and 3-months follow-up
  A 11 item-questionnaire answered on a 7 point likert scale from 1(never) to 7(always)
Changes in Illness perception Measured by the self-report questionnaire Brief Illness perception Questionnaire | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  A questionnaire with 11 items answered on a scale from 0 - 10
Changes in Illness perception rated by parents, measured by the parent-report questionnaire Illness perception regarding child's symptoms Questionnaire | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  A questionnaire with 11 items answered on a scale from 0 - 10
Changes in Illness worry Measured by the self-report questionnaire Childhood Illness Attitude Scale | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The cognitive domain of the questionnaire is used, it consists of 11 items, answers: never, sometimes or always
Changes in Acceptance, measured by the self-report questionnaire Chronic pain Acceptance Questionnaire -adolescents | At baseline, mid-treatment, end-treatment and 3-months follow-up
  Two items from the self-report questionnaire Chronic pain Acceptance Questionnaire -adolescents are used. 2 selected items, answered on a 5-point scale from 0 (never true) to 4 (always true)
Changes in PARENTAL Illness Worry measured by the self-report The Health Anxiety by Proxy Scale (HAPYS) questionnaire | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  Parental illness worry for their child, measured by the self-report The questionnaire covers 26 items about health anxiety by proxy, rated on a five-point scale (from "not at all"/"never" to "a whole lot"/"most of the time"). And five items about the impact of the worries rated on a four-point scale (from "no" to "yes, severely").
Changes in PARENTAL Emotional distress measured by the self-report questionnaire Symptom Check List (SCL-8) | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The questionnaire consist of 8 items answered on a 5 point scale from 0 (not at all) to 4 (a whole lot)
Changes in Adult Response to Child's Symptoms - PARENTS by the self-report questionnaire Adult Response to Children's Symptoms | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  Protect and Monitor scale from the the questionnaire Adult Response to Children's Symptoms used, 15 items answered on a 5 point scale from 0(never) to 4 (always)
Changes in School absence / Work absence parent | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  Question about Hours / Days missed from school/work last month. Parental rated for children aged 8-12 years, self-rated for adolescents aged 13-17 years, self-rated for parents

OTHER OUTCOMES:
Treatment satisfaction by the self-report questionnaire Modified Experience of Service Questionnaire | At 10 weeks of treatment (End of treatment)
  10 items rated either true, partly true, not true or don't know and 3 open end questions about experience of treatment,
Adverse events | At 10 weeks of treatment (End of treatment)
  Open end questions. Parents to children aged 8-12 years will answer on behalf of their children and adolescents aged 13-17 years will answer themselves.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Ulrikka Rask, Professor, MD, PhD, Study Chair — Aarhus University and Aarhus University Hospital, Child and Adolescents Psychiatry
Locations (1):
- Aarhus University and Aarhus University Hospital, Child and Adolescents Psychiatry, Aarhus, Denmark

REFERENCES:
- [Derived] Nielsen ES, Kallesoe K, Lalouni M, Carlsen AH, Frostholm L, Bonnert M, Rask CU. Trajectories of change in pediatric functional abdominal pain disorders during Internet cognitive behavior therapy: A single case experimental study. J Pain. 2025 Jun;31:105407. doi: 10.1016/j.jpain.2025.105407. Epub 2025 Apr 25. PMID 40288508
- [Derived] Skovslund Nielsen E, Kallesoe K, Bennedsen Gehrt T, Bjerre-Nielsen E, Lalouni M, Frostholm L, Bonnert M, Rask CU. Trajectories of Change, Illness Understanding, and Parental Worries in Children and Adolescents Undergoing Internet-Delivered Cognitive-Behavioral Therapy for Functional Abdominal Pain Disorders: Protocol for a Single-Case Design and Explorative Pilot Study. JMIR Res Protoc. 2025 Jan 7;14:e58563. doi: 10.2196/58563. PMID 39773759